CLINICAL TRIAL: NCT00817414
Title: A Phase II, Randomized, Double-blind, Placebo Controlled, Multi-center Study to Evaluate the Effects of LCI699 on Cortisol in Patients With Hypertension
Brief Title: A Study to Evaluate the Effects of LCI699 on Cortisol in Participants With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Great Lakes Drug Development, Inc. (Industry); Integrium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CLCI699A2215; 2008-007337-49 (EudraCT Number)
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Results first posted 2021-06-02 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
Keywords: Blood Pressure; Hypertension; Cortisol
MeSH Terms: conditions — Hypertension | interventions — Osilodrostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: LCI699 0.5 mg QD (Experimental): Participants received LCI699 0.5 mg, capsules, orally, once daily (QD), with or without food for up to 6 weeks.
  Interventions: Drug: LCI699
- Cohort A: LCI699 1.0 mg QD (Experimental): Participants received LCI699 1.0 mg, capsules, orally, QD, with or without food for up to 6 weeks.
  Interventions: Drug: LCI699
- Cohort B1: LCI699 1.0 mg BID (Experimental): Participants received LCI699 1.0 mg, capsules, orally, twice daily (BID), with or without food for up to 6 weeks.
  Interventions: Drug: LCI699
- Cohort B1: LCI699 2.0 mg QD (Experimental): Participants received LCI699 2.0 mg, capsules, orally, QD, with or without food for up to 6 weeks.
  Interventions: Drug: LCI699
- Placebo (Placebo Comparator): Participants received LCI699-matching placebo, capsules, orally, QD or BID, with or without food for up to 6 weeks.
  Interventions: Drug: LCI699-matching placebo

INTERVENTIONS:
Drug: LCI699-matching placebo — LCI699-matching placebo oral capsules
  Arms: Placebo
Drug: LCI699 — LCI699 oral capsules
  Arms: Cohort A: LCI699 0.5 mg QD; Cohort A: LCI699 1.0 mg QD; Cohort B1: LCI699 1.0 mg BID; Cohort B1: LCI699 2.0 mg QD

SUMMARY:
This study determined the maximum dose of LCI6999 with respect to effect on the ACTH-stimulated cortisol response in participants with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension with blood pressure ≥ 140/90 millimeters of mercury (mmHg) and < 180/110 mmHg on current antihypertensive treatment
* Male and female participants 18-75 years of age
* Participants must weigh at least 50 kilograms (kg)

Exclusion Criteria:

* Recent history of myocardial infarction, heart failure, unstable angina, coronary artery bypass graft, percutaneous coronary intervention, hypertensive encephalopathy, cerebral accident or transient ischemic attack
* Clinically significant electrocardiography (ECG) findings related to cardiac conduction defects
* Type 1 diabetes or uncontrolled type 2 diabetes (haemoglobin A1c [HbA1c] > 9%)
* Malignancies within the last 5 years (excluding basal cell skin cancer)
* Liver disease

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-01-14 (Actual); Primary Completion 2009-08-12 (Actual); Study Completion 2009-08-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- United States (10):
  - Impact Clinical Trials, Beverly Hills, California
  - Associated Pharmaceutical Research Center, Inc, Buena Park, California
  - Innovative Clinical Research, Inc, Harbor City, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - Metro Clinical Research, Littleton, Colorado
  - Clinical Study Center of Asheville, LLC, Asheville, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Tipton Medical & Diagnostic Center, Tipton, Pennsylvania
  - Punzi Medical Center, Carrollton, Texas
  - dgd Research, Inc, San Antonio, Texas
- Encode Clinic, Reykjavik, SA, Iceland

REFERENCES:
- [Derived] Schumacher CD, Steele RE, Brunner HR. Aldosterone synthase inhibition for the treatment of hypertension and the derived mechanistic requirements for a new therapeutic strategy. J Hypertens. 2013 Oct;31(10):2085-93. doi: 10.1097/HJH.0b013e328363570c. PMID 24107737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 10 investigative sites in the United States and Iceland from 14 January 2009 to 12 August 2009.
Pre-assignment Details: A total of 63 participants with essential hypertension taking at least one anti-hypertensive treatment were randomized to receive LCI699 in comparison with placebo in an escalated dose design for 6 weeks.
Groups:
- Cohort A: LCI699 1 mg QD: Participants received LCI699 1.0 mg, capsules, orally, QD, with or without food for up to 6 weeks.
- Cohort B1: LCI699 1 mg BID: Participants received LCI699 1.0 mg, capsules, orally, twice daily (BID), with or without food for up to 6 weeks.
- Cohort B1: LCI699 2 mg QD: Participants received LCI699 2.0 mg, capsules, orally, QD, with or without food for up to 6 weeks.
- Placebo: Participants received LCI699-matching placebo, capsules, orally, QD or BID with or without food for up to 6 weeks.
Period: Overall Study
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1 mg QD | Cohort B1: LCI699 1 mg BID | Cohort B1: LCI699 2 mg QD | Placebo
Started | 12 | 12 | 13 | 13 | 13
Completed | 10 | 9 | 9 | 1 | 11
Not Completed | 2 | 3 | 4 | 12 | 2
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0
Not completed — Low Adrenocorticotropic Hormone (ACTH)- Stimulated Cortisol | 0 | 1 | 2 | 4 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 1
Not completed — Dose Arm Exceeds Maximum Tolerated Dose (MTD) | 0 | 0 | 0 | 7 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1 mg QD | Cohort B1: LCI699 1 mg BID | Cohort B1: LCI699 2 mg QD | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 13 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (6.37) | 54.2 (16.01) | 57.9 (9.09) | 56.2 (10.37) | 56.8 (10.08) | 56.3 (10.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 3 | 5 | 4 | 21
  Male | 8 | 7 | 10 | 8 | 9 | 42

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of LCI699 With Respect to Effect on the Adrenocorticotropic Hormone (ACTH)-Stimulated Cortisol Response Following ACTH Stimulation in Hypertensive Participants
Description: As per the protocol, MTD is the dose at which 4 participants exhibited ACTH-stimulated cortisol results <400 nanomoles per liter (nmol/L). The change in the distribution across the treatments were analyzed using 1- way analysis of variance (ANOVA) for continuous variables.
Time Frame: Up to Week 6
Population: Safety set population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number (90% Confidence Interval); unit: milligrams (mg)
Groups:
- LCI699: Participants received LCI699 capsules, orally, QD or BID, with or without food for up to 6 weeks.
Arm/Group | LCI699
Number analyzed (Participants) | 63
milligrams (mg) | 1.30 [0.88 to 1.81]

2. Secondary Outcome: LCI699 Exposure-response Relationship on Cortisol Levels Following ACTH Stimulation in Hypertensive Participants
Description: Exposure-response relationship was assessed using ACTH stimulation test. Tests were done 2 hours after study drug administration (i.e., at peak LCI699 concentrations). An increase in cortisol greater than >500 nmol at 60 minutes after ACTH administration was expected.
Time Frame: Up to Week 6
Population: Safety set population included all participants who were randomized and received at least 1 dose of study drug. Number analyzed is the number of participants with data available for analyses at the given timepoint.
Measure: Mean (Standard Error); unit: nanomoles per liter (nmol/L)
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD | Placebo
Number analyzed (Participants) | 11 | 12 | 12 | 13 | 12
nanomoles per liter (nmol/L)
  Day 7 | 690.0 (32.288) | 669.40 (30.903) | 625.06 (30.965) | 562.04 (30.325) | 799.06 (31.161)
  Day 28: number analyzed (Participants) | 10 | 11 | 12 | 10 | 12
  Day 28 | 634.87 (32.181) | 573.41 (30.642) | 554.79 (29.466) | 539.09 (32.826) | 804.86 (29.786)
  Day 42: number analyzed (Participants) | 8 | 8 | 12 | 7 | 11
  Day 42 | 647.51 (45.593) | 626.08 (45.441) | 539.68 (37.146) | 479.91 (48.865) | 812.91 (39.096)

3. Secondary Outcome: LCI699 Plasma Concentration Post LCI699 Administration at Day 7
Time Frame: Predose and 3 hours post-dose on Day 7
Population: Pharmacokinetic (PK) set population included all participants with sufficient LCI699 plasma samples at post-baseline visits.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 11 | 12 | 13 | 13
nanogram per milliliter (ng/mL) | 1.51 (36) | 2.88 (41) | 3.92 (31) | 6.73 (23)

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of LCI699
Time Frame: Days 7, 28: Pre-dose and 3 hours post-dose; Day 30: Pre-dose; Day 42: Pre-dose and 0.5, 1, 2, 3, 4, and 8-hours post-dose
Population: PK set population included all participants with sufficient LCI699 plasma samples at post-baseline visits. Overall number analysed is the number of participants with data available for these analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 10 | 7 | 12 | 4
ng/mL | 1.42 (36) | 2.94 (35) | 4.62 (35) | 8.86 (21)

5. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of LCI699
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 10 | 7 | 12 | 4
hour (hr) | 2.21 [1.0 to 4.0] | 1.00 [1.0 to 4.0] | 1.00 [0.5 to 4.0] | 1.00 [1.0 to 3.0]

6. Secondary Outcome: Area Under the Concentration Time Curve From Time 0 to 8 Hours Post LCI699 Administration (AUC0-8)
Time Frame: Day 42: Pre-dose and 0.5, 1, 2, 3, 4, and 8-hours post-dose
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 10 | 7 | 12 | 4
nanogram*hour per milliliter (ng*hr/mL) | 6.60 (42) | 14.1 (30) | 24.1 (39) | 46.4 (13)

7. Secondary Outcome: Area Under the Concentration Time Curve Over the Dosing Interval (AUC0-τ) for LCI699
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 9 | 6 | 11 | 4
ng*hr/mL | 9.23 (50) | 18.8 (51) | 30.6 (41) | 68.9 (19)

8. Secondary Outcome: Apparent Terminal Half-life (T1/2) of LCI699
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD
Number analyzed (Participants) | 9 | 6 | 11 | 4
hr | 4.67 (37) | 3.79 (43) | 5.52 (33) | 4.90 (17)

9. Secondary Outcome: Number of Participants With Adverse Event (AEs)
Description: An AE is an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives.
Time Frame: Up to 8 weeks
Population: Safety set population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1 mg QD | Cohort B1: LCI699 1 mg BID | Cohort B1: LCI699 2 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 13
Participants | 6 | 9 | 10 | 10 | 10

10. Secondary Outcome: Percentage of Participants With a Mean Sitting Systolic Blood Pressure (MSSBP) Response and MSSBP Control at Week 6 Last Observation Carried Forward (LOCF), as Measured by Office Blood Pressure (OBP)
Description: Automated arterial BP determinations was made with an automated BP device (such as the Omron BP monitor) in accordance with the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV. Sitting and standing blood pressure (BP) and heart rate (HR) measurements were performed. MSSBP response was defined as the percentage of participants with a MSSBP <140 mmHg or a >=20 mmHg reduction from baseline. MSSBP control was defined as the percentage of participants with a MSSBP <140 mmHg for non-diabetic participants and <130mHg for diabetic participants.
Time Frame: Week 6
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1 mg QD | Cohort B1: LCI699 1 mg BID | Cohort B1: LCI699 2 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 13
percentage of participants
  MSSBP Response | 58.3 | 50.0 | 69.2 | 76.9 | 61.5
  MSSBP Control | 50.0 | 41.7 | 61.5 | 76.9 | 53.8

11. Secondary Outcome: Percentage of Participants With a Mean Sitting Diastolic Blood Pressure (MSDBP) Response and MSDBP Control at Week 6 LOCF, as Measured by OBP
Description: Automated arterial BP determinations was made with an automated BP device (such as the Omron BP monitor) in accordance with the Guidelines for management of hypertension: report of the 4th working party of the British Hypertension Society, 2004-BHS IV. Sitting and standing BP and HR measurements were performed. MSDBP response was defined as the percentage of participants with a MSDBP <90 mmHg or a >= 10 mmHg reduction from baseline. MSDBP control was defined as the percentage of participants with a MSDBP <90 mmHg for non-diabetic participants and <80mHg for diabetic participants.
Time Frame: Week 6
Population: FAS population included all participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1 mg QD | Cohort B1: LCI699 1 mg BID | Cohort B1: LCI699 2 mg QD | Placebo
Number analyzed (Participants) | 12 | 12 | 13 | 13 | 13
percentage of participants
  MSDBP Response | 58.3 | 66.7 | 100 | 76.9 | 61.5
  MSDBP Control | 58.3 | 66.7 | 76.9 | 76.9 | 46.2

ADVERSE EVENTS:
Time Frame: Up to 8 weeks
Description: An AE is an adverse medical event which occurs in a participant of the study and which is not necessarily in a causal relationship with the treatment the participant receives.
Arm/Group | Cohort A: LCI699 0.5 mg QD | Cohort A: LCI699 1.0 mg QD | Cohort B1: LCI699 1.0 mg BID | Cohort B1: LCI699 2.0 mg QD | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/13 | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 6/12 | 9/12 | 10/13 | 10/13 | 10/13
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: LCI699 0.5 mg QD (N=12) | Cohort A: LCI699 1.0 mg QD (N=12) | Cohort B1: LCI699 1.0 mg BID (N=13) | Cohort B1: LCI699 2.0 mg QD (N=13) | Placebo (N=13)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
ACTH stimulation test abnormal (Investigations) | 0 | 1 | 2 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 3 | 0 | 1
Headache (Nervous system disorders) | 1 | 4 | 2 | 2 | 3
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Testicular pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Peripheral coldness (Vascular disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.